CLINICAL TRIAL: NCT03397160
Title: Development, Validation, and Dissemination of an Integrated Risk Prediction Model and Decision Aid to Discern Aggressive Versus Indolent Prostate Cancer
Brief Title: Pioneering Advances in Care and Education (PACE)
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: CentraCare Adult & Pediatric Urology (Unknown); Lancaster Urology (Unknown); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); Palo Alto Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-12951 / UCSF-HDFCC 17553; A-17812.5a,b,c,d,f (Other: HRPO-U.S. Army Medical Research and Materiel Command); NCI-2018-01341 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-11-30; First posted 2018-01-11 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Decision Support Systems, Clinical; Prostate Cancer
Keywords: Prostate cancer; Transformative Impact Award; Early stage; Active surveillance; Decision aid; Coaching session; Personalized; University of California, San Francisco (UCSF); Validation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a site-randomized, cluster-crossover clinical trial of a decision support intervention (DSI) vs. usual care, among men with low prognostic risk prostate cancer, to assess differences in informed decision making (i.e., knowledge), anxiety, and decision quality and self-efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Participants assigned to the control arm will receive usual care, including whatever information materials are provided to them by their urologist.
- Decision Support Intervention (DSI) (Active Comparator): Participants assigned to the intervention will receive Decision Support Intervention in the form of a decision aid plus health coaching. The decision aid (delivered by internet and as a Portable Document Format (PDF) document) provides participants with a report on options and outcomes as described in the literature; along with more tailored risk information. The tailored risk information will include their estimated risk of harboring more aggressive prostate cancer based on their clinical/pathologic features (i.e., "My Clinical Risk"). The DSI was developed and piloted at UCSF according to the International Patient Decision Aid Standards (see http://ipdas.ohri.ca/) (IRS# 14-13332), and incorporates tailored risk models developed and validated.
  Interventions: Behavioral: Decision Support Intervention (DSI)

INTERVENTIONS:
Behavioral: Decision Support Intervention (DSI) — A question list (QL) that includes areas of patient concern are created by the health coach for use by the patient and the urologist at their first consultation visit where they discuss the extent of their cancer and consider treatment options. The coach uses the Prostate Cancer SCOPED model to complete a "Prostate Cancer SCOPED Model Form". The SCOPED model uses concepts such as the situation, choices (treatment), objectives (personal goals and priorities), people (involved in supporting a treatment decision), evaluation and decisions (clarifying which choice is best and next steps).
  Other Names: PCa SCOPED model
  Arms: Decision Support Intervention (DSI)

SUMMARY:
This clinical trial evaluates the use of novel decision support educational materials and services using health coaches. The study includes men newly diagnosed with low-risk prostate cancer. A 160 men will be recruited. Half of the men will receive a call from a health coach before their initial consultation visit with their urologist to review their treatment concerns and questions. The other half will receive usual care provided by the urologist, such as educational materials and services provided by the urologist.

DETAILED DESCRIPTION:
A critical public health need exists for improved prognostic tools to distinguish aggressive from slow growing prostate cancer at diagnosis, and for better support systems to guide patients in decision-making regarding management options.

Decision support interventions that are tailored to specific clinical conditions are known to have increased patient self-efficacy, knowledge, question-asking, and satisfaction; and decreased decisional conflict, regret, anxiety, and distress.

To reduce the risk of over-treatment, our team has developed individual risk prediction models that we have now integrated into our decision support intervention (DSI).

Delivering such decision support intervention should increase patient knowledge and question-asking by the patient to their doctor.

The decision support intervention can be delivered by telephone and or the Internet.

ELIGIBILITY:
Inclusion Criteria:

* Male >=18 years of age and newly diagnosed prostate cancer (PCa) (within 3-months).
* Documentation of a low-risk PCa diagnosis as evidenced by clinical features of the following criteria:

  * PSA test at diagnosis <=15 ng/ml
  * Localized PCa (cT1/T2,N0,M0)
  * Biopsy Gleason grade 2-6 OR (or 3+4 AND <=33% cores are positive for adenocarcinoma)

    ***A minimum of 10 diagnostic cores taken by a systematic directed approach. Sampling may be obtained by target transrectal ultrasound (TRUS) or MRI imaging.
  * No treatment yet

    * No previous radiation or simultaneous use of androgen deprivation
    * Prior use of 5-alpha reductase inhibitor is allowed if they have been stopped for 6 or more months and biopsy performed when patient was not taking the drug
  * English language proficient and ability to provide informed consent
  * Managing urologist considers them a candidate for active surveillance
* Written informed consent (and assent when applicable) obtained from subject and ability for subject to comply with the requirements of the study, including the ability to read and speak English.

Exclusion Criteria:

* Participants will be ineligible if they:

  1. have pursued any active therapy for prostate cancer will be excluded;
  2. are unable to read/speak English; or
  3. if their managing urologist does NOT deem them as a candidate for active surveillance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Decision Quality Index (DQI) scores | 12 months
  The DQI measures patient Knowledge, Concordance, and Decision process. For each fact about prostate cancer item, a correct response = 1 point. Missing responses=0 points. Total score is calculated for all patients who complete at least half of the items and scaled from 0-100%, with higher scores indicating greater knowledge. Patients rate their goals and concerns on an 11-point importance scale from 0 (not important at all) to 10 (extremely important). These questions + one question about patient's treatment preference can be used to calculate a concordance score. Patients are asked about whether they were offered a choice, how much pros and cons were discussed, and whether the health care provider asked for their preferences. Participants get 1 point for a response of "yes" / "a lot/some.", total points are summed, then divided by total number of items for a decision making process score from 0-100%. Higher scores indicate a more shared decision making process.

SECONDARY OUTCOMES:
Memorial Anxiety Scale for Prostate Cancer (MAX-PC) scores | 12 months
  The MAX-PC is an 18-item questionnaire with a 4-point Likert-type scale asking how frequently certain "comments made by men about prostate cancer" were true of the respondent (Roth et al., 2003). Each item is scored from 0 to 4 with anchors ranging from "Not at all" to "Often." The scale can be scored in its entirety by summing all the items or summary scores can be grouped into Prostate Cancer Anxiety (11 items), Prostate-specific antigen (PSA) Anxiety (3 items), or Fear of Re-occurrence (4 items).
Decision Self-Efficacy (DSE) Scores | 12 months
  The DSE measures self-confidence or belief in one's ability to make informed decisions and participate in shared decision making with health professionals. It is a 11-item instrument with a five-point response scale ranging from 0 (not at all confident) to 4 (very confident).

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Carroll, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - Palo Alto Medical Foundation, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - CentraCare Clinic Adult & Pediatric Urology, Sartell, Minnesota
  - Lancaster Urology, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available through a formal data request
URL: https://urology.ucsf.edu/research/cancer/study-proposals-and-working-with-data

REFERENCES:
- [Background] https://www.frontiersin.org/articles/10.3389/fruro.2023.1127089/full
- See also: UCSF Department of Urology - Study Proposals and Working with Data — https://urology.ucsf.edu/research/cancer/study-proposals-and-working-with-data

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT03397160/Prot_SAP_003.pdf
  • Informed Consent Form: 2017: Approved Informed Consent Form (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03397160/ICF_001.pdf
  • Informed Consent Form: 2018: Approved Informed Consent Form (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03397160/ICF_002.pdf